CLINICAL TRIAL: NCT03470467
Title: Posterior Reversible Encephalopathy Syndrome in the Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Ictal Group (Other)
Collaborators: Versailles Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICTAL PRES REGISTRY
Record Dates: First submitted 2018-03-09; First posted 2018-03-20 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Posterior Reversible Encephalopathy Syndrome
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention planed

SUMMARY:
Posterior Reversible Encephalopathy Syndrome prospective (PRES) registry. Data collection using a standardized form : demographic data and data related to the PRES, including circumstances of onset, dates and times of onset and of symptoms control, on-scene clinical findings, clinical and radiological features of PRES, pre-hospital and hospital care providers, timing of antiepileptic, antihypertensive drugs and supportive treatments, results of etiological investigations, cause of PRES, type and dosage of antiepileptic and antihypertensive drugs. Dates and times of EEG monitoring, EEG results, radiological and biological investigations. Outcomes including vital status and Glasgow Outcome Scale score at ICU and hospital discharge, day-90 and 1-year after SE and determined based on data in the ICU and/or neurologist charts and/or patients phone interview

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* Posterior Reversible Encephalopathy Syndrome defined as:

  * combination of consciousness impairment, seizure activity, headaches, visual abnormalities, nausea/vomiting, and focal neurological signs AND
  * cerebral imaging abnormalities involving the white matter (brain CT scan hypodensities AND/OR Brain MRI hypoT1, hyper T2 FLAIR)
* intensive care unit admission

Exclusion Criteria:

* normal cerebral imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: critically ill patients requiring ICU hospitalisation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome | 1 year
  A favorable outcome is defined by a Glasgow Outcome Scale (GOS) of 5. The Glasgow Outcome Scale (GOS) will be determined during a structured interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]

SECONDARY OUTCOMES:
Favorable outcome | 3-months and 5-years, 10-years
  A favorable outcome is defined by a Glasgow Outcome Scale (GOS) of 5. The Glasgow Outcome Scale (GOS) will be determined during a structured interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]
Functional impairment | 3-months and 1-year, 5-years, 10-years
  Percentages of patients with functional impairments (motor, sensitive or cognitive deficits)
Low or moderate disability | 3-months and 1-year, 5-years, 10-years
  Low or moderate disability is defined by a Glasgow Outcome Scale (GOS) of 4 or 5.
  The Glasgow Outcome Scale (GOS) will be determined during a structured interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]
Recurrent PRES | 3-months and 1-year, 5-years, 10-years
  percentages of the patients that experience recurrence of PRES [defined as a variable combination of consciousness impairment, seizure activity, headaches, visual abnormalities, nausea/vomiting, and focal neurological signs AND cerebral imaging abnormalities involving the white matter (brain CT scan hypodensities AND/OR Brain MRI hypoT1, hyper T2 FLAIR)]
Mortality rate | ICU, hospital discharge, 3-months and 1-year, 5-years, 10-years
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LEGRIEL, MD, Principal Investigator — Ictal Group
Locations (1):
- Intensive Care Unit - Versailles Hospital, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Undecided